CLINICAL TRIAL: NCT04792398
Title: Effects of Botulinum Toxin Type A (Xeomin®) Injections Into Bilateral Masseter Muscles for Management of Bruxism and Associated Symptoms: Single Center Open Label Longitudinal Pilot Study
Brief Title: Bruxism Xeomin® Intervention Trial
Acronym: BRUX-XIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dominik Ettlin (Other)
Collaborators: Merz Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Dominik Ettlin, Study Principal Investigator, MD, DMD, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRUX-XIT
Record Dates: First submitted 2021-03-02; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Sleep Bruxism, Adult
MeSH Terms: conditions — Sleep Bruxism | interventions — incobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: Observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sleep Bruxism Subjects (Experimental): Ultrasound guided BTX-A injection: 25 units (divided in two injections) in each masseter muscle.
  One-time intervention. Effect observation by measuring various biosignals (EMG, EOG, EEG), bite force, chewing efficiency, psychometric assessments.
  Interventions: Drug: Incobotulinumtoxin A (BTX A) Xeomin®

INTERVENTIONS:
Drug: Incobotulinumtoxin A (BTX A) Xeomin® — Injections into the masseter muscles bilaterally (25 Units per muscle applied with 2 injections in each muscle)

SUMMARY:
The purpose of this study is to test whether severe masticatory muscle spasms during sleep (e.g. teeth clenching and grinding, known as "bruxism" in technical jargon) demonstrably decrease after application of botulinum toxin type A (Xeomin®). Xeomin® has so far been used to relieve spasms of other muscles and is an approved drug in Switzerland. This study is now intended to test the suitability of this drug for relaxation of the masseter muscle.

DETAILED DESCRIPTION:
Bruxism is a prevalent condition that differentially burdens individuals. The overall objective of this pilot study is to measure the effects of BTX-A (Xeomin®) injections into bilateral masseter muscles for the management of sleep bruxism and associated symptoms. The hypothesis is that BTX-A reduces masticatory muscle activity. The aim of this study is to instrumentally monitor subjects closely over an extended time period of three months before and after application of BTX-A.

Botulinum toxin type A ( BTX A; Xeomin ® ) temporarily blocks neuromuscular synapses. It is successfully and safely used therapeutically in various types of movement disorders and in chronic migraineurs. The mechanism of action of this treatment is related to a reduction of neurotransmitter release leading to reduced muscle activity.

The following Null hypothesis will be tested:

Injections of Xeomin® into the masseter muscles bilaterally (25 Units per muscle applied with 2 injections in each muscle) have no effect on bruxism measured by A) Masticatory muscle activity (1° objective) B) Subjects' well-being (2° objective) C) Sensitivity of masticatory muscles and jaw joints (2° objective) D) Anxiety over tooth wear (2° objective) E) Disturbed sleep by bed partner (2° objective)

Following instruments will be used:

1. WISE questionnaires. A comprehensive web-based interdisciplinary symptom evaluation tool.
2. Algometer for sensitivity measure of masticatory muscles and jaw joints.
3. Bio-signal recorder. Parallel to the Electromyography (EMG) of the masseter muscles, other bio-signals such as a number of electroencephalographic (EEG) derivations, electrooculogram (EOG ) as well as an electrocardiogram (ECG) will be recorded, in order to detect sleep stages and better identify bruxism episodes. The device used in this study has been approved for projects NIH #2R01DE016417-05A1 and #1 R01DE028548-01.
4. Ultrasound for masseter muscle thickness measure
5. Dual-color chewing gum for chewing efficiency measure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years;
* patients complaining of bruxism and/or bruxism-related symptoms.
* Sufficient knowledge of German to understand the patient information and the trial arrangement.

Exclusion Criteria:

* Contraindications for Xeomin® treatment such as generalized disorders of muscle activity (myasthenia gravis, Lambert-Eaton-Rooke syndrome);
* documented hypersensitivity to one of the components,
* local infection of the injection sites;
* intake of anticoagulants or muscle relaxing medications;
* recreational drugs.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change of maximum EMG amplitudes | days 1-14, days 29-42
  Change of average of maximum EMG amplitudes of all bruxism events per night between days 1-14 (baseline) and days 29-42.
Verbal Rating Scale of Global impression of change | day 154
  Verbal Rating Scale (VRS) containing the following levels "much worse", "slightly worse", "no change", "slightly improved", "much improved" of "global impression of change" at the end of the study (day 154)

SECONDARY OUTCOMES:
Change of maximum EMG amplitude | days 1-14, days 15-28, days 85-98, days 141-154
  Change of average of maximum EMG amplitudes of all bruxism events per night between days 1-14 (baseline) and days 15-28, 85-98, and 141-154.
EMG amplitude at maximum voluntary contraction | days 1-14, days 15-28, days 85-98, days 141-154
  EMG signal amplitude (RMS) at maximum voluntary contraction (MVC) in [V]
number of masseter contraction episodes per hour (N/h) | days 1-14, days 15-28, days 85-98, days 141-154
  number of masseter contraction episodes per hour calculated from EMG signal amplitude normalized on MVC [N/h]
duration of masseter contraction episodes (Dur) | days 1-14, days 15-28, days 85-98, days 141-154
  duration of masseter contraction episodes in [sec] calculated from EMG signal amplitude normalized on MVC
EMG-Index | days 1-14, days 15-28, days 85-98, days 141-154
  EMG-Index = 0.5 x N/h + Dur
EMG Duty Factor | days 1-14, days 15-28, days 85-98, days 141-154
  EMG duty factor = % duration of muscle activity/total recording time
Sensitivity of masticatory muscles and jaw joints | day 1, 14, 28, 42, 98, 154
  Sensitivity of masticatory muscles and jaw joints in [N]
Self-report of bruxism | day 1, 14, 28, 42, 98, 154
  Yes/No answer to direct question
Numerical Rating Scale masseter muscle pain | day 1, 14, 28, 42, 98, 154
  Numerical Rating Scale (NRS) (0-10) with 0 = no pain and 10 = worst imaginable pain
Numerical Rating Scale report of spontaneous facial pain | day 1, 14, 28, 42, 98, 154
  Numerical Rating Scale (NRS) (0-10) with 0 = no pain and 10 = worst imaginable pain
Numerical Rating Scale report of jaw movement related facial pain | day 1, 14, 28, 42, 98, 154
  Numerical Rating Scale (NRS) (0- 10) with 0 = no pain and 10 = worst imaginable pain
Numerical Rating Scale report of anxiety over tooth wear | day 1, 14, 28, 42, 98, 154
  Numerical Rating Scale (NRS) (0-10) with 0 = no anxiety and 10 = worst imaginable anxiety
Numerical Rating Scale disturbed sleep of bed partner | day 1, 14, 28, 42, 98, 154
  Numerical Rating Scale (NRS) (0-10) with 0 = no disturbed sleep and 10 = worst imaginable sleep

CONTACTS AND LOCATIONS:
Overall Officials: Dominik A Ettlin, MD, DMD, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Center of Dental Medicine, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ettlin DA, Sommer I, Bronnimann B, Maffioletti S, Scheidt J, Hou MY, Lukic N, Steiger B. Design, construction, and technical implementation of a web-based interdisciplinary symptom evaluation (WISE) - a heuristic proposal for orofacial pain and temporomandibular disorders. J Headache Pain. 2016 Dec;17(1):77. doi: 10.1186/s10194-016-0670-5. Epub 2016 Aug 31. PMID 27581159
- [Background] Iwasaki LR, Gonzalez YM, Liu H, Marx DB, Gallo LM, Nickel JC. A pilot study of ambulatory masticatory muscle activities in temporomandibular joint disorders diagnostic groups. Orthod Craniofac Res. 2015 Apr;18 Suppl 1(0 1):146-55. doi: 10.1111/ocr.12085. PMID 25865543
- [Background] Silva LC, Nogueira TE, Rios LF, Schimmel M, Leles CR. Reliability of a two-colour chewing gum test to assess masticatory performance in complete denture wearers. J Oral Rehabil. 2018 Apr;45(4):301-307. doi: 10.1111/joor.12609. Epub 2018 Feb 9. PMID 29356092
- See also: Homepage Company used Medical Device Algomed — http://www.cephalon.eu/products/sensory/algomed/